CLINICAL TRIAL: NCT05689749
Title: Evaluation of Lacrimal Gland Involvement by Superb Microvascular Imaging Ultrasonography Technique in Patients With Sjögren Syndrome
Brief Title: Superb Microvascular Imaging Ultrasonography of Lacrimal Gland in Patients With Sjögren Syndrome
Acronym: SMI
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Ender Salbaş, Physical Medicine & Rehabilitation Specialist, MD, Nigde Omer Halisdemir University
Other Study IDs: ES02
Record Dates: First submitted 2022-12-28; First posted 2023-01-19 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Inflammation; Sjogren's Syndrome; Gland; Inflammation
Keywords: superb microvascular imaging; microvascularization; Sjogren's syndrome; disease activitiy
MeSH Terms: conditions — Inflammation; Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with Sjögren's syndrome: Participants with the diagnose of Sjögren's syndrome; Patients with a confirmed diagnosis who are being followed and treated by a rheumatologist.
  Interventions: Device: Superb Microvascular Imaging (SMI) (Toshiba)
- Volunteers who has not dry eye complaints and Sjögren's syndrome diagnosis.: Voluntary participants without any rheumatic disease diagnosis, without Sjögren's syndrome diagnosis, without dry eye complaints will constitute the other group.
  Interventions: Device: Superb Microvascular Imaging (SMI) (Toshiba)

INTERVENTIONS:
Device: Superb Microvascular Imaging (SMI) (Toshiba) — To determine whether SMI has diagnostic value for detecting the inflammatory state in the lacrimal glands in Sjögren's syndrome and whether it has any superiority compared to Power Doppler and Color Doppler modalities.

SUMMARY:
A prospective study will be conducted to evaluate inflammatory activity in lacrimal glands due to Sjögren's syndrome on Superb Microvascular Imaging (SMI), gray scale ultrasound (US), color Doppler US and Power Doppler US.

DETAILED DESCRIPTION:
In the disease activity index recommended by EULAR, the European Rheumatology Association, to evaluate the disease activity of patients with Sjögren's syndrome, it is recommended to measure the swelling in the gland by performing a clinical examination for glandular activity. However, it is not practical to measure the size of these glands due to their location.

In studies in which lacrimal glands were evaluated by ultrasonographic methods, parameters such as gland size measurement, gland heterogeneity and Doppler activity were reported to be very successful in differentiating patients from healthy controls.

Determining the presence and characteristics of vascular flow is an important part of ultrasonographic examinations. However, small vessels and low velocities are not always possible to detect with conventional color and power Doppler ultrasound. Sonographic examination will be inconclusive, especially if the presence of vascular flow or activity needs to be addressed as a basis for diagnosis and follow-up. Superb Microvascular Imaging (SMI) is a new vascular imaging mode that provides low speed and visualization of microvascular flow. SMI uses an algorithm that can suppress parasitic reverberations to extract flow signals and displays this information as a color overlay image or a monochromatic or color flow map.There are studies that report that Superb Microvascular Imaging (SMI), a new and up-to-date Ultrasonography technology, is more sensitive in detecting the activity of Rheumatic diseases. In this respect, there are no studies evaluating the inflammatory activity of lacrimal glands with SMI method.

Therefore, a prospective study will be conducted to evaluate the inflammation detecting performance of SMI, gray scale US, color Doppler US and Power Doppler US. The null hypothesis that there is no difference between Doppler US and SMI methods in the detection of increased inflammatory activity in Sjögren's syndrome patients.

ELIGIBILITY:
For the first group:

Inclusion Criteria:

* Patients diagnosed with Sjögren's syndrome
* Age between 18-65

Exclusion Criteria:

* History of eye or face trauma or surgery
* Diabetes mellitus
* Pregnancy

For the second group:

Inclusion Criteria:

* asymptomatic eye (no dry eye or dry mouth),
* no previous trauma or surgery on face or eye,
* no history of systemic inflammatory disorders.

Exclusion Criteria:

* History of eye or face trauma or surgery
* Diabetes mellitus
* Pregnancy
* Rheumatological diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients who diagnosed as Sjögren's syndrome as the first group.
  * Healthy participants as the second group
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Schirmer's test | 1 year
  The tip of a special paper strip is placed inside the lower eyelid of each eye. During the test on both eyes, the eyes are asked to remain closed for 5 minutes. After 5 minutes the doctor removes the paper and measures how much is moistened.
Ocular Surface Disease Index (OSDI) | 1 year
  Participants will be asked to answer a 12-question questionnaire asking about various conditions and symptoms related to dry eye.It is a 12-item questionnaire designed to provide a rapid assessment of the symptoms of ocular irritation consistent with dry eye disease and their impact on vision-related functioning. The 12 items of the OSDI questionnaire were graded on a scale of 0 to 4, where 0 indicates none of the time; 1, some of the time; 2, half of the time; 3, most of the time; and 4, all of the time. The total OSDI score was then calculated on the basis of the following formula: OSDI=[(sum of scores for all questions answered) × 100]/[(total number of questions answered) × 4].
McMonnies Dry Eye Questionnaire | 1 year
  Participants will be asked to answer a 12-question questionnaire asking about various conditions and symptoms related to dry eye. It is presented on a single page and includes 12 questions that focus on clinical risk factors for DES. The questions employ polytomous response options that vary in number and type. For example, question 1 has three response categories consisting of yes (2), no (0), and uncertain (1), whereas question 9 has four response categories, consisting of never (0), sometimes (1), often (2), and constantly (3).
Ultrasonographic Evaluation; Superb Microvascular Imaging, GrayScale Imaging, Color Doppler Imaging, Power Doppler Imaging | 1 year
  Four-stage classify will be use for grading these images; Grade 0: No vascularity in lacrimal and parotid gland, Grade 1: One or two focal color-encoded spots in lacrimal and parotid gland, Grade 2: One linear color-encoded line or more than two focal colorencoded spots in lacrimal and parotid gland, Grade 3: More than one linear color-encoded line in lacrimal and parotid gland

CONTACTS AND LOCATIONS:
Overall Officials: Ender Salbas, MD, Study Director — Nigde Omer Halisdemir University
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Turkey (Türkiye)